CLINICAL TRIAL: NCT06139887
Title: Examining a Strategy to Engage Rural Veteran Patients After Community Care Treatment
Brief Title: Suicide Prevention Program for Veterans Discharged From Community Care Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: White River Junction Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: VHA Office of Rural Health (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1701666
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Results first posted 2025-08-22 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Suicide Prevention
Keywords: Mental health education; Clinical trial; Suicidal ideation; Suicide, attempted
MeSH Terms: conditions — Suicide Prevention; Suicidal Ideation; Suicide, Attempted | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two groups in parallel: BESST plus standard care vs. standard care alone.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will be blinded to treatment allocation and will remind the participant at each contact to not disclose their treatment status.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BESST (Experimental): Patients randomized to the BESST intervention arm will receive the BESST intervention combined with standard mental health care.
  Interventions: Behavioral: BESST; Other: Standard Mental Health Care
- Control (Other): Patients randomized to the control arm will receive standard mental health care alone.
  Interventions: Other: Standard Mental Health Care

INTERVENTIONS:
Behavioral: BESST — The BESST intervention is a suicide prevention program designed to meet the unique needs of Veterans receiving care from community mental health treatment settings. BESST can be delivered by a trained mental health staff member, such as a mental health nurse, social worker, psychologist, or psychiatrist. The intervention consists of two synergistic components that work to support the patient after a mental health-related discharge in community settings: 1) Brief educational session, where the patient receives a one-hour, one-on-one, personalized educational session on suicide prevention; 2) Seven regular contacts after discharge, where the study interventionist who delivered the brief educational visit will contact the patient to monitor the patient's symptoms, assess treatment adherence, review their safety plan, and assist the patient with engaging in care, if needed.
  Arms: BESST
Other: Standard Mental Health Care — Patients randomized to the control arm will receive standard mental health care alone. Standard mental health care simply refers to the regular care provided to patients around the time of discharge from community care settings.
  Other Names: Standard Care

SUMMARY:
The goal of this pilot randomized controlled trial is to test an adapted suicide prevention program (the Building VA Engagement, Self-efficacy, and Social Support To Prevent Suicide or BESST) in rural Veterans discharged from community care mental health treatment settings. The main question it aims to answer is:

* Does BESST combined with standard care improve suicide-related outcomes among this population compared to standard care alone?

Participants will be assigned by change to a treatment group. Some will receive the BESST intervention combined with standard care, and some will receive standard care alone. All participants will be in this research study for up to three months.

Those receiving the BESST intervention will have:

* 1 one-hour brief educational session;
* Seven follow-up check-ins (~30 minutes each)

All participants will have three assessment interviews where they will be asked about their mental health and treatment received outside of the VA.

The investigators will compare participants assigned to the BESST intervention combined with standard care vs participants assigned to standard care alone to see if the BESST intervention improves suicide-related outcomes.

ELIGIBILITY:
Inclusion Criteria:

* The patient was recently discharged from a VA community care mental health treatment setting
* The patient is at risk for self-harm
* Be a patient connected to the White River Junction VA Medical Center (VAMC), the Togus VA Medical Center (VAMC), or the Manchester VA Medical Center (VAMC);
* Be a Veteran;
* Be 18 years or older;
* Be able to speak English;

Exclusion Criteria:

* Unable to provide informed consent;
* The investigators do not plan to enroll any potentially vulnerable populations including prisoners, institutionalized patients, or involuntarily committed patients;
* Study physician deems the patient not clinically appropriate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-04-17 (Actual); Study Completion 2025-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Riblet, MD, MPH, Principal Investigator — White River Junction VA Medical Center
Locations (1):
- White River Junction VA Medical Center, White River Junction, Vermont, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BESST | Control
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BESST | Control | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.7 (9.08) | 42.0 (11.63) | 42.35 (10.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 9 | 9 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 9 | 10 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 10 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 10 | 20
The Beck Scale for Suicidal Ideation (BSS) [Mean (Standard Deviation); unit: units on a scale] — The BSS ranges from 0-38. While there is no established BSS cutoff score to classify risk of suicide, there is some evidence that higher scores on the BSS correspond to more severe suicidal ideation and that a change of five points or more on the total BSS scores may be of clinical relevance. Mean BSS scores at baseline were calculated.
  units on a scale | 4.6 (6.293) | 9.4 (9.8) | 7.0 (8.39)
The Beck Scale for Hopelessness (BHS) [Mean (Standard Deviation); unit: units on a scale] — The BHS ranges from 0-20 with higher scores associated with worse hopelessness. The mean BHS scores at baseline were calculated.
  units on a scale | 9.8 (4.49) | 8.7 (3.43) | 9.25 (3.93)
Interpersonal Needs Questionnaire-15, Perceived Burdensomeness (INQ-15 PB) [Mean (Standard Deviation); unit: units on a scale] — The INQ-15 is a 15-item self-report scale that assesses thwarted belongingness (9 items) and perceived burdensomeness (6 items). Each item on the INQ-15 is measured on a 7-point Likert scale, with higher scores indicating lower perceived connectedness. The score range for the entire INQ-15 scale is 15-105, with the score range for perceived burdensomeness being 6-42. The perceived burdensomeness mean scores on the INQ-15 at baseline were calculated.
  units on a scale | 16.2 (8.65) | 15.3 (6.82) | 15.75 (7.59)
Interpersonal Needs Questionnaire-15, Thwarted Belongingness (INQ-15 TB) [Mean (Standard Deviation); unit: units on a scale] — The INQ-15 is a 15-item self-report scale that measures thwarted belongingness (9 items) and perceived burdensomeness (6 items). Each item on the INQ-15 is measured on a 7-point Likert scale, with higher scores indicating lower perceived connectedness. The score range for the entire INQ-15 scale is 15-105, with the score range for thwarted belongingness being 7-63. Mean thwarted belonging scores on the INQ-15 at baseline were calculated.
  units on a scale | 34.2 (10.62) | 31.3 (7.54) | 32.75 (9.09)
The Multidimensional Scale of Perceived Social Support (MSPSS) [Mean (Standard Deviation); unit: units on a scale] — The MSPSS is a 12-item self-reported scale that is designed to inquire about support from several sources including family, friends, and significant others. The MSPSS scale has been shown to have good internal and test-retest reliability as well as good validity. The score range is 1-7 with higher values indicating increased perception of social support. The mean MSPSS scores at baseline were calculated.
  units on a scale | 4.34 (1.45) | 4.99 (0.84) | 4.67 (1.20)
Suicide Related Coping Scale (SRCS) External Coping Subscale [Mean (Standard Deviation); unit: units on a scale] — This scale includes 17 questions related to a patient's perception of their ability to cope with their suicidal thoughts. Each item is assessed using a 5-point Likert scale. The scale includes two subscales including an External Coping subscale and an Internal Coping Subscale. The score range for the entire scale is 0-68 with the External Coping being 0-28. Higher scores indicate increased perception of suicide-related external coping. Mean scores at baseline were calculated.
  units on a scale | 22.0 (4.42) | 23.4 (3.66) | 22.7 (4.01)
Suicide Related Coping Scale (SRCS) Internal Coping Subscale [Mean (Standard Deviation); unit: units on a scale] — This scale includes 17 questions related to a patient's perception of their ability to cope with their suicidal thoughts. Each item is assessed using a 5-point Likert scale. The SRCS scale includes two subscales including an External Coping subscale and an Internal Coping Subscale. The score range for the entire scale is 0-68 with the Internal Coping being 0-28. Higher scores indicate increased perception of suicide-related internal coping. Mean scores at baseline were calculated.
  units on a scale | 18.4 (6.79) | 20.0 (5.56) | 19.2 (6.09)
Generalized Self-Efficacy Scale (GES) [Mean (Standard Deviation); unit: units on a scale] — The General Self-Efficacy Scale (GSES) is a valid scale of self-efficacy that is designed for the general population (12 years or older) and it has been tested in various countries. It is a 10-item psychometric scale that is designed to assess optimistic self-beliefs to cope with a variety of difficult demands in life. Total scores range from 10 to 40, with higher scores suggesting increased self-efficacy.
  units on a scale | 27.0 (6.02) | 25.9 (4.41) | 26.45 (5.17)

OUTCOME MEASURES:

1. Primary Outcome: Suicidal Ideation: The Beck Scale for Suicidal Ideation (BSS)
Description: The Beck Scale for Suicidal Ideation (BSS) ranges from 0-38. While there is no established BSS cutoff score to classify suicide risk, there is evidence that higher scores on the BSS correspond to more severe suicidal ideation and that a change of five points or more on the total BSS scores may be clinically relevant.
Time Frame: 3 months post-baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BESST | Control
Number analyzed (Participants) | 10 | 10
units on a scale | 2.0 (4.22) | 10.7 (9.48)

2. Secondary Outcome: Hopelessness: Beck Hopelessness Scale (BHS)
Description: The Beck Hopelessness Scale (BHS) is a 20-item self-report scale that assesses hopelessness over the past seven days. Patients report on feelings about the future, loss of motivation, and future expectations. Total scores range from 0 to 20, with higher scores suggesting more hopelessness. The BHS has good reliability and validity and is sensitive to change. There is some evidence that the BHS may be a measure of risk of suicide.
Time Frame: 3 months post-baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BESST | Control
Number analyzed (Participants) | 10 | 10
units on a scale | 5.6 (4.74) | 10.4 (6.50)

3. Secondary Outcome: Connectedness: Interpersonal Needs Questionnaire-15 (INQ-15) Perceived Burdensomeness
Description: The Interpersonal Needs Questionnaire-15 (INQ-15) is a 15-item self-report scale that measures thwarted belongingness (9 items) and perceived burdensomeness (6 items). Each item is measured on a 7-point Likert scale, with higher scores suggesting lower perceived connectedness. The score range for the entire scale is 15-105, with the score range for perceived burdensomeness being 6-42.
Time Frame: 3 months post-baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BESST | Control
Number analyzed (Participants) | 10 | 10
units on a scale | 10.2 (5.98) | 17.4 (12.24)

4. Secondary Outcome: Connectedness: Interpersonal Needs Questionnaire-15 (INQ-15) Thwarted Belongingness
Description: The Interpersonal Needs Questionnaire-15 (INQ-15) is a 15-item self-report scale that measures thwarted belongingness (9 items) and perceived burdensomeness (6 items). Each item is measured on a 7-point Likert scale, with higher scores suggesting lower perceived connectedness. The score range for the entire scale is 15-105, with the score range for thwarted belongingness being 7-63.
Time Frame: 3 months post-baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BESST | Control
Number analyzed (Participants) | 10 | 10
units on a scale | 29.1 (11.3) | 32.3 (15.72)

5. Secondary Outcome: Patient Engagement: General Self-Efficacy Scale (GSES)
Description: The General Self-Efficacy Scale (GSES) is a valid scale of self-efficacy that is designed for the general population (12 years or older) and it has been tested in various countries. It is a 10-item psychometric scale that is designed to assess optimistic self-beliefs to cope with a variety of difficult demands in life. Total scores range from 10 to 40, with higher scores suggesting increased self-efficacy.
Time Frame: 3 months post-baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BESST | Control
Number analyzed (Participants) | 10 | 10
units on a scale | 30.4 (7.85) | 28.1 (6.59)

6. Secondary Outcome: Patient Engagement: Suicide-Related Coping Scale (SRCS) External Coping Subscale
Description: The Suicide-Related Coping Scale (SRCS) includes 17 questions related to a patient's perception of their ability to cope with suicidal thoughts. Each item is assessed using a 5-point Likert scale. The scale includes two subscales including an External Coping subscale and an Internal Coping Subscale. The score range for the entire scale is 0-68 with the External Coping being 0-28 and the Internal Coping being 0-28. Higher scores indicate increased perception of suicide-related coping.
Time Frame: 3 months post-baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BESST | Control
Number analyzed (Participants) | 10 | 10
units on a scale | 24.6 (3.63) | 22.1 (7.26)

7. Secondary Outcome: Patient Engagement: Suicide Related Coping Scale (SRCS) Internal Coping Subscale
Description: as for outcome 6
Time Frame: 3 months post-baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BESST | Control
Number analyzed (Participants) | 10 | 10
units on a scale | 25.2 (4.39) | 20.2 (7.79)

8. Secondary Outcome: Number of Participants With Suicide Attempts
Description: Suicide attempts is measured using the seven-item subscale on the Columbia-Suicide Severity Rating Scale (C-SSRS), a valid and reliable scale that asks patients to self-report on suicide attempts.
Time Frame: 3 months post-baseline
Measure: Count of Participants; unit: Participants
Arm/Group | BESST | Control
Number analyzed (Participants) | 10 | 10
Participants | 0 | 0

9. Secondary Outcome: Number of Participants With Substance Use at 3 Months Post-baseline
Description: The investigators will assess substance use at follow-up assessments using a timeline follow-back approach. This method is commonly used in research studies to assess substance use patterns. Numerical scores do not apply to this assessment.
Time Frame: 3 months post-baseline
Measure: Count of Participants; unit: Participants
Arm/Group | BESST | Control
Number analyzed (Participants) | 10 | 10
Participants | 3 | 5

ADVERSE EVENTS:
Time Frame: Adverse event data were collected throughout the entirety of the study participant activities (approximately 3 months).
Description: Because our study enrolled a high-risk group of patients, it was expected that patients would potentially report worsening mental health symptoms and/or problems specific to substance use. In some of these cases, the patients would then be expected to be hospitalized or treated in the emergency room for these reasons. Based on local approval from our institutional review board, we treated these events as adverse events.
Arm/Group | BESST | Control
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 4/10 | 4/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BESST (N=10) | Control (N=10)
Suicidal behavior (Psychiatric disorders) | 2 (2) | 4 (4) — Suicidal behavior including worsening suicidal ideation or preparatory behaviors. We determined that these symptoms or behaviors were expected in the population and unrelated to study procedures.
Psychological distress (Psychiatric disorders) | 2 (2) | 0 (0) — Self report of increased psychological distress. We determined that these symptoms were expected in the population and unrelated to study procedures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-11-27): https://cdn.clinicaltrials.gov/large-docs/87/NCT06139887/Prot_SAP_001.pdf
  • Informed Consent Form (2024-01-02): https://cdn.clinicaltrials.gov/large-docs/87/NCT06139887/ICF_000.pdf